CLINICAL TRIAL: NCT00374582
Title: End Stage Liver Disease and Body Composition Assessment: Utilizing Bioelectric Impedance Analysis (BIA)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cincinnati (Other)
Responsible Party: Guy Neff, MD, University of Cincinnati
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BIA
Record Dates: First submitted 2006-09-08; First posted 2006-09-11 (Estimated); Last update posted 2011-03-04 (Estimated); Status verified 2011-03

CONDITIONS: End Stage Liver Disease
Keywords: Bioelectric impedance analysis; BIA; ESLD; LVP; Large volume paracentesis; Ascites; Liver; Hepatic
MeSH Terms: conditions — End Stage Liver Disease; Ascites

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Bodystat Quadscan 4000 — device determining body composition and nutritional status
Device: bodystat quadscan 400 — device determining body composition and nutritional status

SUMMARY:
The purpose of this research study is to see how effective bioelectric impedance analysis (BIA) is in determining body composition (the amount of fat versus muscle in the body) and nutritional status in patients with End Stage Liver Disease (ESLD)

DETAILED DESCRIPTION:
The aim of this study is to report the validity of mBIA to determine body composition changes pre and post LVP (Large Volume Paracentesis)

* 18 years of age or older
* Cirrhotic patients with refractory ascites requiring LVP (a treatment to remove large volumes of excess fluid from the abdominal cavity)
* End Stage Liver Disease

ELIGIBILITY:
Inclusion Criteria:

* Patients with ESLD requiring LVP.
* Age over 18.
* Ability to provide written informed consent.

Exclusion Criteria:

* Organ retransplant candidates.
* Patient with use of any investigational agent within 30 days before LVP.
* Pregnant or lactating.
* Patients with non-bioprosthetic heart valves pacemakers, defibrillators, artificial joints, pins, plates, or other types of metal objects in the body.
* Amputations other than fingers or toes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2006-09; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Efficacy and utility of BIA in determining body composition and nutritional status using multi-frequency machines in patients with ESLD and ascites requiring LVP. | Before and after large volume paracentesis

SECONDARY OUTCOMES:
Quantify the difference in BIA pre and post LVP to evaluate the impact of oncotic pressure in the assessment of total body composition. | Before and after large volume paracentis

CONTACTS AND LOCATIONS:
Overall Officials: Guy Neff, MD, Principal Investigator — University of Cincinnati
Locations (1):
- University of Cincinnati, Cincinnati, Ohio, United States